CLINICAL TRIAL: NCT06729632
Title: Non-Invasive System to Deliver Therapeutic Hypothermia for Protection Against Noise-Induced Hearing Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Restorear Devices LLC (Industry)
Collaborators: University of Miami (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DC018760; 2R44DC018760-02A1 (NIH)
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Noise Exposure; Noise-induced Hearing Loss; Noise; Adverse Effect; Mild Therapeutic Hypothermia; Cooling; Occupational Exposure; Occupational Health; Hidden Hearing Loss
Keywords: hearing preservation; hearing loss; noise-induced hearing loss; noise exposure; mild therapeutic hypothermia; cooling; post-exposure; prevention
MeSH Terms: conditions — Hearing Loss, Noise-Induced; Hearing Loss, Hidden; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Aim 1 studies will use a crossover study design. Aim 2 studies will use a parallel model.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Safety Arm (Experimental): Non-firefighter control subjects will receive MTH-treatment and normothermia-sham through the device alternated over 8 sessions. Subjective assessments and audiologic testing pre- and post-treatments will be compared between MTH-treatment and sham in each subject. n=24.
  Interventions: Device: Cold pack-delivered mild therapeutic hypothermia
- Efficacy Arm 1 - Treatment (Experimental): Firefighters will receive hypothermia treatment delivered with ReBound devices, applied post-work shift. Baseline hearing function will be measured prior to initiation of the treatment. Treatments and functional assessments will be repeated quarterly over one year. Temporary and permanent threshold changes in this chronically noise exposed group of firefighters receiving MTH-treatment will be compared with firefighters receiving sham-treatment and with controls receiving MTH-treatment. Subjects in this group will also be sent home with a device to use after noise exposure during the study period. They will complete weekly, remote surveys collecting data on their noise exposure and device use. n=24.
  Interventions: Device: Cold pack-delivered mild therapeutic hypothermia
- Efficacy Arm 2 - Non-Therapeutic (No Intervention): Firefighters will receive non-therapeutic "treatment" delivered with normothermic ReBound devices, applied post-work shift. Baseline hearing function will be measured prior to initiation of the treatment. Treatments and functional assessments will be repeated quarterly over one year. n=24.
- Efficacy Arm 3 - Control (Active Comparator): Age- and sex-matched non-firefighter control group will receive MTH-treatment quarterly over the same duration. Baseline hearing function will be measured prior to initiation of the treatment. Treatments and functional assessments will be repeated quarterly over one year. Subjects in this group will also be sent home with a device to use after noise exposure during the study period. They will complete weekly, remote surveys collecting data on their noise exposure and device use. n=24.
  Interventions: Device: Cold pack-delivered mild therapeutic hypothermia

INTERVENTIONS:
Device: Cold pack-delivered mild therapeutic hypothermia — Mild therapeutic hypothermia (cooling), delivered non-invasively to the structures of the inner ear (cochlea) for 30 minutes, using headband-style proprietary device, ReBoundRx.
  Arms: Efficacy Arm 1 - Treatment; Efficacy Arm 3 - Control; Safety Arm

SUMMARY:
The goal of this interventional clinical study is to investigate the use of mild therapeutic hypothermia devices for preservation of sensory structures in the cochlea after noise exposure. The main aims of the study are:

1. To test the safety and best duration for use for a new hypothermia device.
2. To determine if the hypothermia device helps decrease noise-induced hearing loss in a group of firefighters.

Participants will wear the mild therapeutic hypothermia therapy devices immediately after a fire service shift serially over a year. Researchers will compare results from those receiving the therapy to those from a control group (individuals receiving no therapy and a sham therapy).

DETAILED DESCRIPTION:
Noise-induced hearing loss (NIHL) is highly prevalent among occupationally at-risk service groups like the military and firefighters, with disabilities that result in significant healthcare burden, negatively impacting performance on duty and quality of life. Exposure to noise can cause permanent threshold shifts (PTS) with accompanying hair cell loss, or temporary threshold shifts (TTS), with no evident hair cell loss. Noise exposure can also result in rapid and permanent loss of synaptic elements and cochlear nerve terminals with irreversible hearing impairment and long-term degeneration of spiral ganglion (SG) cell bodies.

Currently no FDA-approved treatments are available to prevent or treat NIHL. Delivering pharmaceutical compounds over time, identification of safe dosages, and a critical timeframe relative to noise-exposure remain clinically challenging. RestorEar Devices LLC has developed a non-pharmaceutical application of mild therapeutic hypothermia (MTH) to protect residual sensory structures and function of the cochlea. MTH is a proven and well-established therapy for neuroprotection. This approach for MTH application is based on significant prior and on-going research that highlights its utility for residual hearing preservation against cochlear implant surgical trauma, ototoxicity, and noise exposure. With SBIR Phase I support, the investigators have successfully demonstrated that effective non-invasive, non-pharmaceutical therapeutic hypothermia can be delivered to the inner ear sensory structures. The investigators have built, calibrated, and tested ReBoundTM, a headband with cooling gel packs placed in contact with the surface of the mastoid. ReBoundTM delivers MTH safely and repeatedly for up to 30 minutes. In this study, the investigators aim to extend this application to human subjects and test safety and efficacy against NIHL in noise-exposed firefighters and matched controls with the collaboration of researchers at the University of Miami.

Aim 1: Evaluate safety of MTH with ReBoundTM devices. With the first in-human studies, the investigators aim to show that MTH can be safely delivered to the inner ear using ReBound. In a randomized study, non-firefighter control subjects will receive MTH-treatment and normothermia-sham (non-cooled gel pack) through the device alternated over 8 sessions. Subjective assessments and audiologic testing (pure tone audiometry, auditory brainstem responses, distortion product otoacoustic emissions and electrocochleography) pre- and post-treatments will be compared between MTH-treatment and sham in each subject. Results of Aim 1 will support the hypothesis that this approach will deliver therapeutic hypothermia to the cochleae and that repeated application will not negatively affect hearing function in healthy subjects.

Aim 2: Validate efficacy of the ReBoundTM MTH devices for mitigating NIHL in an occupationally at-risk group. Based on strong preliminary results, the investigators hypothesize that acute application of MTH in noise-exposed firefighters will reduce temporary changes in auditory function. Firefighters will be divided equally into two treatment groups, MTH-treatment and normothermia-sham. These treatments will be delivered with ReBound, with and without cooled gel packs, applied post-duty. MTH-treatment will also be applied in an age- and sex-matched control group over the same duration. Baseline hearing function will be measured prior to initiation of the treatment. Treatments and the functional assessments will be repeated quarterly over one year. Temporary and permanent threshold changes in this chronically the noise exposed group of firefighters receiving MTH-treatment will be compared with firefighters receiving sham-treatment and with controls receiving MTH-treatment. MTH-groups will also be sent home with a ReBound band and instructed to use it after noise exposure. Subjective assessments will be sent weekly to these groups to evaluate the use pattern of the device. Results of these studies will firmly establish MTH for mitigating NIHL.

This research will be highly impactful given the significant adverse effects of NIHL, an unmet clinical need, and the high translational potential of MTH for mitigating NIHL.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 years old at the time of signing the consent form
* Fluency in English

Exclusion Criteria:

* Abnormal tympanometric findings
* Abnormal pure tone audiometry from 500-8,000 Hz (Non-firefighters only)
* Significant history of noise exposure (Non-firefighters only)
* Temporomandibular joint disorder
* Otologic pathologies (including, but not limited to): acoustic neuroma/vestibular schwannoma, chronic ear disease, Meniere's disease, documented fluctuating hearing loss, or ototoxicity
* Current recipients of medical, pharmacologic, or therapeutic intervention for tinnitus or other otologic conditions
* Active hearing aid users
* Adults unable to consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pure Tone Audiometry | Safety Arm: Twice per week, pre- and post- treatment, to the end of treatment at 4 weeks. Efficacy Arms: Every 3 months, pre- and post-treatment, for 1 year.
  Pure Tone Audiometry (PTA) will be performed in the Safety and Efficacy arms immediately post-treatment. PTA will be performed at baseline and immediately post-treatment in the Safety Arm, 8 times over 4 weeks. In the Efficacy Arms, it will be completed quarterly before and immediately post-treatment.
Distortion Product Otoacoustic Emissions | Safety Arm: Twice per week, pre- and post- treatment, to the end of treatment at 4 weeks. Efficacy Arms: Every 3 months, pre- and post-treatment, for 1 year.
  Distortion Product Otoacoustic Emissions (DPOAE) will be performed in the Safety and Efficacy Arms immediately post-treatment. DPOAE will be performed at baseline and immediately post-treatment in the Safety Arm, 8 times over 4 weeks. In the Efficacy Arms, it will be completed quarterly before and immediately post-treatment.
Adverse Event Questionnaire | Immediately post-treatment; 3-hours and 24-hours post-treatment.
  The 2 question Adverse Event Questionnaire (AEQ) will be administered in both the Safety and Efficacy Arms. It will collect data on any adverse event associated with use of the device.

SECONDARY OUTCOMES:
Device Acceptance Questionnaire | Safety Arm: Post-initial treatment and at the end of week 4 post-enrollment; Efficacy Arms: Post-initial treatment and at the end of 12 months
  11 question survey about subjective experience and acceptance of the treatment. Includes Likert Scale questions about comfort, likelihood of use of the device, etc.
Weekly Use Surveys | Weekly, from enrollment to end of treatment at 52 weeks.
  Experimental Efficacy Arm and Non-Firefighter Control Arms for Efficacy Study will complete weekly, 3 question survey monitoring the use of the device at home. Firefighters will be asked how many shifts they had that week and how many times they used the device. Non-firefighters will be asked about their noise exposure and device use.

CONTACTS AND LOCATIONS:
Overall Officials: Suhrud M Rajguru, PhD, Principal Investigator — RestorEar Devices
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Presneill J, Gantner D, Nichol A, McArthur C, Forbes A, Kasza J, Trapani T, Murray L, Bernard S, Cameron P, Capellier G, Huet O, Newby L, Rashford S, Rosenfeld JV, Smith T, Stephenson M, Varma D, Vallance S, Walker T, Webb S, James Cooper D; POLAR investigators and the ANZICS Clinical Trials Group. Statistical analysis plan for the POLAR-RCT: The Prophylactic hypOthermia trial to Lessen trAumatic bRain injury-Randomised Controlled Trial. Trials. 2018 Apr 27;19(1):259. doi: 10.1186/s13063-018-2610-y. PMID 29703266
- [Background] Hospital, R., Randomized Controlled Trial of Long-term Mild Hypothermia for Severe Traumatic Brain Injury (LTH-Ⅰ), in ClinicalTrials.gov. 2017: https://www.clinicaltrials.gov/ct2/show/NCT01886222.
- [Background] Azman, A.S. and R.L. Hudak, An evaluation of sound restoration hearing protection devices and audibility issues in mining. Noise Control Engineering Journal, 2011. 59(6): p. 622-630
- [Background] Rabinowitz, P.M., The Public Health Significance of Noise-Induced Hearing Loss, in Noise-Induced Hearing Loss: Scientific Advances, C.G. LePrell, et al., Editors. 2012. p. 13-25.
- [Background] Nadon, V. and J. Voix, Effects of noise exposure on hearing health evaluated through short interval otoacoustic emission monitoring: Preliminary results with low and moderate noise exposure groups. The Journal of the Acoustical Society of America, 2018. 144(3): p. 1789-1789
- [Background] Thepaksorn, P., et al., Occupational hazard exposures and health risks at wooden toys industry in Southern Thailand. Human and Ecological Risk Assessment, 2020. 26(8): p. 2162-2172
- [Background] Emara, A. and T. Gabr, Chronic noise exposure: impact on the vestibular function. Advanced Arab Academy of Audio-Vestibulogy Journal, 2014. 1(2): p. 71-79
- [Background] Humes LE, J.L., Durch JS, Noise and military service: implications for hearing loss and tinnitus. Washington, DC: Institute of Medicine of the National Academies, 2005
- [Background] Basner M, Babisch W, Davis A, Brink M, Clark C, Janssen S, Stansfeld S. Auditory and non-auditory effects of noise on health. Lancet. 2014 Apr 12;383(9925):1325-1332. doi: 10.1016/S0140-6736(13)61613-X. Epub 2013 Oct 30. PMID 24183105
- [Background] Hawkins JE Jr, Johnsson LG, Stebbins WC, Moody DB, Coombs SL. Hearing loss and cochlear pathology in monkeys after noise exposure. Acta Otolaryngol. 1976 Mar-Apr;81(3-4):337-43. doi: 10.3109/00016487609119971. PMID 817561
- [Background] Kujawa SG, Liberman MC. Synaptopathy in the noise-exposed and aging cochlea: Primary neural degeneration in acquired sensorineural hearing loss. Hear Res. 2015 Dec;330(Pt B):191-9. doi: 10.1016/j.heares.2015.02.009. Epub 2015 Mar 11. PMID 25769437
- [Background] Fernandez KA, Jeffers PW, Lall K, Liberman MC, Kujawa SG. Aging after noise exposure: acceleration of cochlear synaptopathy in "recovered" ears. J Neurosci. 2015 May 13;35(19):7509-20. doi: 10.1523/JNEUROSCI.5138-14.2015. PMID 25972177
- [Background] Yankaskas K. Prelude: noise-induced tinnitus and hearing loss in the military. Hear Res. 2013 Jan;295:3-8. doi: 10.1016/j.heares.2012.04.016. Epub 2012 May 2. PMID 22575206
- [Background] Liberman MC, Epstein MJ, Cleveland SS, Wang H, Maison SF. Toward a Differential Diagnosis of Hidden Hearing Loss in Humans. PLoS One. 2016 Sep 12;11(9):e0162726. doi: 10.1371/journal.pone.0162726. eCollection 2016. PMID 27618300
- [Background] Valderrama JT, Beach EF, Yeend I, Sharma M, Van Dun B, Dillon H. Effects of lifetime noise exposure on the middle-age human auditory brainstem response, tinnitus and speech-in-noise intelligibility. Hear Res. 2018 Aug;365:36-48. doi: 10.1016/j.heares.2018.06.003. Epub 2018 Jun 12. PMID 29913342
- [Background] Schaette R, McAlpine D. Tinnitus with a normal audiogram: physiological evidence for hidden hearing loss and computational model. J Neurosci. 2011 Sep 21;31(38):13452-7. doi: 10.1523/JNEUROSCI.2156-11.2011. PMID 21940438
- [Background] Perez E, Viziano A, Al-Zaghal Z, Telischi FF, Sangaletti R, Jiang W, Dietrich WD, King C, Hoffer ME, Rajguru SM. Anatomical Correlates and Surgical Considerations for Localized Therapeutic Hypothermia Application in Cochlear Implantation Surgery. Otol Neurotol. 2019 Oct;40(9):1167-1177. doi: 10.1097/MAO.0000000000002373. PMID 31318786
- [Background] Dietrich WD, Bramlett HM. Therapeutic hypothermia and targeted temperature management for traumatic brain injury: Experimental and clinical experience. Brain Circ. 2017 Oct-Dec;3(4):186-198. doi: 10.4103/bc.bc_28_17. Epub 2017 Dec 29. PMID 30276324
- [Background] Alva N, Palomeque J, Carbonell T. Oxidative stress and antioxidant activity in hypothermia and rewarming: can RONS modulate the beneficial effects of therapeutic hypothermia? Oxid Med Cell Longev. 2013;2013:957054. doi: 10.1155/2013/957054. Epub 2013 Dec 2. PMID 24363826
- [Background] Woo JI, Kil SH, Oh S, Lee YJ, Park R, Lim DJ, Moon SK. IL-10/HMOX1 signaling modulates cochlear inflammation via negative regulation of MCP-1/CCL2 expression in cochlear fibrocytes. J Immunol. 2015 Apr 15;194(8):3953-61. doi: 10.4049/jimmunol.1402751. Epub 2015 Mar 16. PMID 25780042
- [Background] Yang WP, Henderson D, Hu BH, Nicotera TM. Quantitative analysis of apoptotic and necrotic outer hair cells after exposure to different levels of continuous noise. Hear Res. 2004 Oct;196(1-2):69-76. doi: 10.1016/j.heares.2004.04.015. PMID 15464303
- [Background] Valero MD, Burton JA, Hauser SN, Hackett TA, Ramachandran R, Liberman MC. Noise-induced cochlear synaptopathy in rhesus monkeys (Macaca mulatta). Hear Res. 2017 Sep;353:213-223. doi: 10.1016/j.heares.2017.07.003. Epub 2017 Jul 8. PMID 28712672
- [Background] Hickman TT, Smalt C, Bobrow J, Quatieri T, Liberman MC. Blast-induced cochlear synaptopathy in chinchillas. Sci Rep. 2018 Jul 16;8(1):10740. doi: 10.1038/s41598-018-28924-7. PMID 30013117
- [Background] Robles L, Ruggero MA. Mechanics of the mammalian cochlea. Physiol Rev. 2001 Jul;81(3):1305-52. doi: 10.1152/physrev.2001.81.3.1305. PMID 11427697
- [Background] Tamames I, King C, Huang CY, Telischi FF, Hoffer ME, Rajguru SM. Theoretical Evaluation and Experimental Validation of Localized Therapeutic Hypothermia Application to Preserve Residual Hearing After Cochlear Implantation. Ear Hear. 2018 Jul/Aug;39(4):712-719. doi: 10.1097/AUD.0000000000000529. PMID 29240567
- [Background] Dugan EA, Bennett C, Tamames I, Dietrich WD, King CS, Prasad A, Rajguru SM. Therapeutic hypothermia reduces cortical inflammation associated with utah array implants. J Neural Eng. 2020 Apr 29;17(2):026035. doi: 10.1088/1741-2552/ab85d2. PMID 32240985
- [Background] Dietrich WD, Levi AD, Wang M, Green BA. Hypothermic treatment for acute spinal cord injury. Neurotherapeutics. 2011 Apr;8(2):229-39. doi: 10.1007/s13311-011-0035-3. PMID 21416406
- [Background] Truettner JS, Bramlett HM, Dietrich WD. Posttraumatic therapeutic hypothermia alters microglial and macrophage polarization toward a beneficial phenotype. J Cereb Blood Flow Metab. 2017 Aug;37(8):2952-2962. doi: 10.1177/0271678X16680003. Epub 2016 Jan 1. PMID 27864465
- [Background] Lotocki G, de Rivero Vaccari JP, Perez ER, Sanchez-Molano J, Furones-Alonso O, Bramlett HM, Dietrich WD. Alterations in blood-brain barrier permeability to large and small molecules and leukocyte accumulation after traumatic brain injury: effects of post-traumatic hypothermia. J Neurotrauma. 2009 Jul;26(7):1123-34. doi: 10.1089/neu.2008.0802. PMID 19558276
- [Background] Purdy PD, Novakovic RL, Giles BP, Miller SL, Riegel MS. Spinal cord hypothermia without systemic hypothermia. AJNR Am J Neuroradiol. 2013 Jan;34(1):252-6. doi: 10.3174/ajnr.A3175. Epub 2012 Jul 5. PMID 22766669
- [Background] Dietrich WD, Bramlett HM. The evidence for hypothermia as a neuroprotectant in traumatic brain injury. Neurotherapeutics. 2010 Jan;7(1):43-50. doi: 10.1016/j.nurt.2009.10.015. PMID 20129496
- [Background] Dietrich WD, Atkins CM, Bramlett HM. Protection in animal models of brain and spinal cord injury with mild to moderate hypothermia. J Neurotrauma. 2009 Mar;26(3):301-12. doi: 10.1089/neu.2008.0806. PMID 19245308
- [Background] Sewell WF, Borenstein JT, Chen Z, Fiering J, Handzel O, Holmboe M, Kim ES, Kujawa SG, McKenna MJ, Mescher MM, Murphy B, Swan EE, Peppi M, Tao S. Development of a microfluidics-based intracochlear drug delivery device. Audiol Neurootol. 2009;14(6):411-22. doi: 10.1159/000241898. Epub 2009 Nov 16. PMID 19923811
- [Background] Gao X, Tao Y, Lamas V, Huang M, Yeh WH, Pan B, Hu YJ, Hu JH, Thompson DB, Shu Y, Li Y, Wang H, Yang S, Xu Q, Polley DB, Liberman MC, Kong WJ, Holt JR, Chen ZY, Liu DR. Treatment of autosomal dominant hearing loss by in vivo delivery of genome editing agents. Nature. 2018 Jan 11;553(7687):217-221. doi: 10.1038/nature25164. Epub 2017 Dec 20. PMID 29258297
- [Background] Kempfle JS, Luu NC, Petrillo M, Al-Asad R, Zhang A, Edge ASB. Lin28 reprograms inner ear glia to a neuronal fate. Stem Cells. 2020 Jul;38(7):890-903. doi: 10.1002/stem.3181. Epub 2020 Apr 30. PMID 32246510
- [Background] Nourbakhsh A, Colbert BM, Nisenbaum E, El-Amraoui A, Dykxhoorn DM, Koehler KR, Chen ZY, Liu XZ. Stem Cells and Gene Therapy in Progressive Hearing Loss: the State of the Art. J Assoc Res Otolaryngol. 2021 Apr;22(2):95-105. doi: 10.1007/s10162-020-00781-0. Epub 2021 Jan 28. PMID 33507440
- [Background] Greenberg JM, Lumbreras V, Pelaez D, Rajguru SM, Cheung HS. Neural Crest Stem Cells Can Differentiate to a Cardiomyogenic Lineage with an Ability to Contract in Response to Pulsed Infrared Stimulation. Tissue Eng Part C Methods. 2016 Oct;22(10):982-990. doi: 10.1089/ten.tec.2016.0232. PMID 28192031
- [Background] Bas E, Van De Water TR, Lumbreras V, Rajguru S, Goss G, Hare JM, Goldstein BJ. Adult human nasal mesenchymal-like stem cells restore cochlear spiral ganglion neurons after experimental lesion. Stem Cells Dev. 2014 Mar 1;23(5):502-14. doi: 10.1089/scd.2013.0274. Epub 2013 Dec 4. PMID 24172073
- [Background] Chen J, Yuan H, Talaska AE, Hill K, Sha SH. Increased Sensitivity to Noise-Induced Hearing Loss by Blockade of Endogenous PI3K/Akt Signaling. J Assoc Res Otolaryngol. 2015 Jun;16(3):347-56. doi: 10.1007/s10162-015-0508-x. Epub 2015 Mar 20. PMID 25790950
- [Background] Batinic-Haberle I, Reboucas JS, Spasojevic I. Superoxide dismutase mimics: chemistry, pharmacology, and therapeutic potential. Antioxid Redox Signal. 2010 Sep 15;13(6):877-918. doi: 10.1089/ars.2009.2876. PMID 20095865
- [Background] Gao G, Liu Y, Zhou CH, Jiang P, Sun JJ. Solid lipid nanoparticles loaded with edaravone for inner ear protection after noise exposure. Chin Med J (Engl). 2015 Jan 20;128(2):203-9. doi: 10.4103/0366-6999.149202. PMID 25591563
- [Background] Bottger EC, Schacht J. The mitochondrion: a perpetrator of acquired hearing loss. Hear Res. 2013 Sep;303:12-9. doi: 10.1016/j.heares.2013.01.006. Epub 2013 Jan 27. PMID 23361190
- [Background] Mukherjea D, Ghosh S, Bhatta P, Sheth S, Tupal S, Borse V, Brozoski T, Sheehan KE, Rybak LP, Ramkumar V. Early investigational drugs for hearing loss. Expert Opin Investig Drugs. 2015 Feb;24(2):201-17. doi: 10.1517/13543784.2015.960076. Epub 2014 Sep 22. PMID 25243609
- [Background] Le Prell CG, Yamashita D, Minami SB, Yamasoba T, Miller JM. Mechanisms of noise-induced hearing loss indicate multiple methods of prevention. Hear Res. 2007 Apr;226(1-2):22-43. doi: 10.1016/j.heares.2006.10.006. Epub 2006 Dec 4. PMID 17141991
- [Background] Kujawa SG, Liberman MC. Translating animal models to human therapeutics in noise-induced and age-related hearing loss. Hear Res. 2019 Jun;377:44-52. doi: 10.1016/j.heares.2019.03.003. Epub 2019 Mar 15. PMID 30903954
- [Background] Bielefeld EC, Kobel MJ. Advances and Challenges in Pharmaceutical Therapies to Prevent and Repair Cochlear Injuries From Noise. Front Cell Neurosci. 2019 Jun 26;13:285. doi: 10.3389/fncel.2019.00285. eCollection 2019. PMID 31297051
- [Background] Hickox AE, Larsen E, Heinz MG, Shinobu L, Whitton JP. Translational issues in cochlear synaptopathy. Hear Res. 2017 Jun;349:164-171. doi: 10.1016/j.heares.2016.12.010. Epub 2017 Jan 7. PMID 28069376
- [Background] Hu N, Rutherford MA, Green SH. Protection of cochlear synapses from noise-induced excitotoxic trauma by blockade of Ca2+-permeable AMPA receptors. Proc Natl Acad Sci U S A. 2020 Feb 18;117(7):3828-3838. doi: 10.1073/pnas.1914247117. Epub 2020 Feb 3. PMID 32015128
- [Background] Xiong H, Long H, Pan S, Lai R, Wang X, Zhu Y, Hill K, Fang Q, Zheng Y, Sha SH. Inhibition of Histone Methyltransferase G9a Attenuates Noise-Induced Cochlear Synaptopathy and Hearing Loss. J Assoc Res Otolaryngol. 2019 Jun;20(3):217-232. doi: 10.1007/s10162-019-00714-6. Epub 2019 Feb 1. PMID 30710318
- [Background] Szobota S, Mathur PD, Siegel S, Black K, Saragovi HU, Foster AC. BDNF, NT-3 and Trk receptor agonist monoclonal antibodies promote neuron survival, neurite extension, and synapse restoration in rat cochlea ex vivo models relevant for hidden hearing loss. PLoS One. 2019 Oct 31;14(10):e0224022. doi: 10.1371/journal.pone.0224022. eCollection 2019. PMID 31671109
- [Background] Hashimoto K, Hickman TT, Suzuki J, Ji L, Kohrman DC, Corfas G, Liberman MC. Protection from noise-induced cochlear synaptopathy by virally mediated overexpression of NT3. Sci Rep. 2019 Oct 25;9(1):15362. doi: 10.1038/s41598-019-51724-6. PMID 31653916
- [Background] Zhang J, Song YL, Tian KY, Qiu JH. Minocycline attenuates noise-induced hearing loss in rats. Neurosci Lett. 2017 Feb 3;639:31-35. doi: 10.1016/j.neulet.2016.12.039. Epub 2016 Dec 19. PMID 28007648
- [Background] Yu Y, Hu B, Bao J, Mulvany J, Bielefeld E, Harrison RT, Neton SA, Thirumala P, Chen Y, Lei D, Qiu Z, Zheng Q, Ren J, Perez-Flores MC, Yamoah EN, Salehi P. Otoprotective Effects of Stephania tetrandra S. Moore Herb Isolate against Acoustic Trauma. J Assoc Res Otolaryngol. 2018 Dec;19(6):653-668. doi: 10.1007/s10162-018-00690-3. Epub 2018 Sep 5. PMID 30187298
- [Background] Someya S, Yu W, Hallows WC, Xu J, Vann JM, Leeuwenburgh C, Tanokura M, Denu JM, Prolla TA. Sirt3 mediates reduction of oxidative damage and prevention of age-related hearing loss under caloric restriction. Cell. 2010 Nov 24;143(5):802-12. doi: 10.1016/j.cell.2010.10.002. PMID 21094524
- [Background] Richter CP, Young H, Richter SV, Smith-Bronstein V, Stock SR, Xiao X, Soriano C, Whitlon DS. Fluvastatin protects cochleae from damage by high-level noise. Sci Rep. 2018 Feb 14;8(1):3033. doi: 10.1038/s41598-018-21336-7. PMID 29445111
- [Background] Campbell KC, Meech RP, Klemens JJ, Gerberi MT, Dyrstad SS, Larsen DL, Mitchell DL, El-Azizi M, Verhulst SJ, Hughes LF. Prevention of noise- and drug-induced hearing loss with D-methionine. Hear Res. 2007 Apr;226(1-2):92-103. doi: 10.1016/j.heares.2006.11.012. Epub 2007 Jan 16. PMID 17224251
- [Background] Bao J, Hungerford M, Luxmore R, Ding D, Qiu Z, Lei D, Yang A, Liang R, Ohlemiller KK. Prophylactic and therapeutic functions of drug combinations against noise-induced hearing loss. Hear Res. 2013 Oct;304:33-40. doi: 10.1016/j.heares.2013.06.004. Epub 2013 Jun 18. PMID 23792074
- [Background] Bas E, Goncalves S, Adams M, Dinh CT, Bas JM, Van De Water TR, Eshraghi AA. Spiral ganglion cells and macrophages initiate neuro-inflammation and scarring following cochlear implantation. Front Cell Neurosci. 2015 Aug 12;9:303. doi: 10.3389/fncel.2015.00303. eCollection 2015. PMID 26321909
- [Background] Tanaka C, Nguyen-Huynh A, Loera K, Stark G, Reiss L. Factors associated with hearing loss in a normal-hearing guinea pig model of Hybrid cochlear implants. Hear Res. 2014 Oct;316:82-93. doi: 10.1016/j.heares.2014.07.011. Epub 2014 Aug 14. PMID 25128626
- [Background] Reiss LA, Stark G, Nguyen-Huynh AT, Spear KA, Zhang H, Tanaka C, Li H. Morphological correlates of hearing loss after cochlear implantation and electro-acoustic stimulation in a hearing-impaired Guinea pig model. Hear Res. 2015 Sep;327:163-74. doi: 10.1016/j.heares.2015.06.007. Epub 2015 Jun 16. PMID 26087114
- [Background] McCullagh MC, Banerjee T, Yang JJ, Bernick J, Duffy S, Redman R. Gender differences in use of hearing protection devices among farm operators. Noise Health. 2016 Nov-Dec;18(85):368-375. doi: 10.4103/1463-1741.195803. PMID 27991469
- [Background] Wu PZ, Liberman LD, Bennett K, de Gruttola V, O'Malley JT, Liberman MC. Primary Neural Degeneration in the Human Cochlea: Evidence for Hidden Hearing Loss in the Aging Ear. Neuroscience. 2019 May 21;407:8-20. doi: 10.1016/j.neuroscience.2018.07.053. Epub 2018 Aug 10. PMID 30099118
- [Background] Le Prell CG, Hammill TL, Murphy WJ. Noise-induced hearing loss: Translating risk from animal models to real-world environments. J Acoust Soc Am. 2019 Nov;146(5):3646. doi: 10.1121/1.5133385. PMID 31795692
- [Background] Tikka C, Verbeek JH, Kateman E, Morata TC, Dreschler WA, Ferrite S. Interventions to prevent occupational noise-induced hearing loss. Cochrane Database Syst Rev. 2017 Jul 7;7(7):CD006396. doi: 10.1002/14651858.CD006396.pub4. PMID 28685503
- [Background] Tessier-Sherman B, Galusha D, Cantley LF, Cullen MR, Rabinowitz PM, Neitzel RL. Occupational noise exposure and risk of hypertension in an industrial workforce. Am J Ind Med. 2017 Dec;60(12):1031-1038. doi: 10.1002/ajim.22775. Epub 2017 Sep 22. PMID 28940215
- [Background] Staudt AM, Whitworth KW, Chien LC, Whitehead LW, Gimeno Ruiz de Porras D. Association of organic solvents and occupational noise on hearing loss and tinnitus among adults in the U.S., 1999-2004. Int Arch Occup Environ Health. 2019 Apr;92(3):403-413. doi: 10.1007/s00420-019-01419-2. Epub 2019 Feb 26. PMID 30806784
- [Background] Sayler SK, Roberts BJ, Manning MA, Sun K, Neitzel RL. Patterns and trends in OSHA occupational noise exposure measurements from 1979 to 2013. Occup Environ Med. 2019 Feb;76(2):118-124. doi: 10.1136/oemed-2018-105041. Epub 2018 Nov 27. PMID 30482879
- [Background] McTague MF, Galusha D, Dixon-Ernst C, Kirsche SR, Slade MD, Cullen MR, Rabinowitz PM. Impact of daily noise exposure monitoring on occupational noise exposures in manufacturing workers. Int J Audiol. 2013 Feb;52 Suppl 1(0 1):S3-8. doi: 10.3109/14992027.2012.743047. PMID 23373740
- [Background] Lie A, Skogstad M, Johannessen HA, Tynes T, Mehlum IS, Nordby KC, Engdahl B, Tambs K. Occupational noise exposure and hearing: a systematic review. Int Arch Occup Environ Health. 2016 Apr;89(3):351-72. doi: 10.1007/s00420-015-1083-5. Epub 2015 Aug 7. PMID 26249711
- [Background] Li X, Dong Q, Wang B, Song H, Wang S, Zhu B. The Influence of Occupational Noise Exposure on Cardiovascular and Hearing Conditions among Industrial Workers. Sci Rep. 2019 Aug 8;9(1):11524. doi: 10.1038/s41598-019-47901-2. PMID 31395914
- [Background] Dzhambov A, Dimitrova D. Occupational Noise Exposure and the Risk for Work-Related Injury: A Systematic Review and Meta-analysis. Ann Work Expo Health. 2017 Nov 10;61(9):1037-1053. doi: 10.1093/annweh/wxx078. PMID 29136415
- [Background] Zhang C, Frye MD, Sun W, Sharma A, Manohar S, Salvi R, Hu BH. New insights on repeated acoustic injury: Augmentation of cochlear susceptibility and inflammatory reaction resultant of prior acoustic injury. Hear Res. 2020 Aug;393:107996. doi: 10.1016/j.heares.2020.107996. Epub 2020 May 18. PMID 32534268
- [Background] Si S, Lewkowski K, Fritschi L, Heyworth J, Liew D, Li I. Productivity Burden of Occupational Noise-Induced Hearing Loss in Australia: A Life Table Modelling Study. Int J Environ Res Public Health. 2020 Jun 29;17(13):4667. doi: 10.3390/ijerph17134667. PMID 32610505
- [Background] Liberman MC, Kujawa SG. Cochlear synaptopathy in acquired sensorineural hearing loss: Manifestations and mechanisms. Hear Res. 2017 Jun;349:138-147. doi: 10.1016/j.heares.2017.01.003. Epub 2017 Jan 10. PMID 28087419
- [Background] Hoffer ME, Balaban C, Slade MD, Tsao JW, Hoffer B. Amelioration of acute sequelae of blast induced mild traumatic brain injury by N-acetyl cysteine: a double-blind, placebo controlled study. PLoS One. 2013;8(1):e54163. doi: 10.1371/journal.pone.0054163. Epub 2013 Jan 23. PMID 23372680
- [Background] Viola P, Scarpa A, Pisani D, Petrolo C, Aragona T, Spadera L, De Luca P, Gioacchini FM, Ralli M, Cassandro E, Cassandro C, Chiarella G. Sub-Clinical Effects of Chronic Noise Exposure on Vestibular System. Transl Med UniSa. 2020 May 31;22:19-23. eCollection 2020 May. PMID 32523903
- [Background] Stewart CE, Kanicki AC, Altschuler RA, King WM. Vestibular short-latency evoked potential abolished by low-frequency noise exposure in rats. J Neurophysiol. 2018 Feb 1;119(2):662-667. doi: 10.1152/jn.00668.2017. Epub 2017 Nov 8. PMID 29118200
- [Background] Stewart CE, Holt AG, Altschuler RA, Cacace AT, Hall CD, Murnane OD, King WM, Akin FW. Effects of Noise Exposure on the Vestibular System: A Systematic Review. Front Neurol. 2020 Nov 25;11:593919. doi: 10.3389/fneur.2020.593919. eCollection 2020. PMID 33324332
- [Background] Stewart C, Yu Y, Huang J, Maklad A, Tang X, Allison J, Mustain W, Zhou W, Zhu H. Effects of high intensity noise on the vestibular system in rats. Hear Res. 2016 May;335:118-127. doi: 10.1016/j.heares.2016.03.002. Epub 2016 Mar 10. PMID 26970474
- [Background] Lien S, Dickman JD. Vestibular Injury After Low-Intensity Blast Exposure. Front Neurol. 2018 May 14;9:297. doi: 10.3389/fneur.2018.00297. eCollection 2018. PMID 29867715
- [Background] Golz A, Westerman ST, Westerman LM, Goldenberg D, Netzer A, Wiedmyer T, Fradis M, Joachims HZ. The effects of noise on the vestibular system. Am J Otolaryngol. 2001 May-Jun;22(3):190-6. doi: 10.1053/ajot.2001.23428. PMID 11351289
- [Background] Ewert DL, Lu J, Li W, Du X, Floyd R, Kopke R. Antioxidant treatment reduces blast-induced cochlear damage and hearing loss. Hear Res. 2012 Mar;285(1-2):29-39. doi: 10.1016/j.heares.2012.01.013. Epub 2012 Feb 6. PMID 22326291
- [Background] Cho SI, Gao SS, Xia A, Wang R, Salles FT, Raphael PD, Abaya H, Wachtel J, Baek J, Jacobs D, Rasband MN, Oghalai JS. Mechanisms of hearing loss after blast injury to the ear. PLoS One. 2013 Jul 1;8(7):e67618. doi: 10.1371/journal.pone.0067618. Print 2013. PMID 23840874
- [Background] Fausti SA, Wilmington DJ, Gallun FJ, Myers PJ, Henry JA. Auditory and vestibular dysfunction associated with blast-related traumatic brain injury. J Rehabil Res Dev. 2009;46(6):797-810. doi: 10.1682/jrrd.2008.09.0118. PMID 20104403
- [Background] Huddle MG, Goman AM, Kernizan FC, Foley DM, Price C, Frick KD, Lin FR. The Economic Impact of Adult Hearing Loss: A Systematic Review. JAMA Otolaryngol Head Neck Surg. 2017 Oct 1;143(10):1040-1048. doi: 10.1001/jamaoto.2017.1243. PMID 28796850
- [Background] Carroll YI, Eichwald J, Scinicariello F, Hoffman HJ, Deitchman S, Radke MS, Themann CL, Breysse P. Vital Signs: Noise-Induced Hearing Loss Among Adults - United States 2011-2012. MMWR Morb Mortal Wkly Rep. 2017 Feb 10;66(5):139-144. doi: 10.15585/mmwr.mm6605e3. PMID 28182600
- [Background] Zhao F, Manchaiah VK, French D, Price SM. Music exposure and hearing disorders: an overview. Int J Audiol. 2010 Jan;49(1):54-64. doi: 10.3109/14992020903202520. PMID 20001447
- [Background] Stucken EZ, Hong RS. Noise-induced hearing loss: an occupational medicine perspective. Curr Opin Otolaryngol Head Neck Surg. 2014 Oct;22(5):388-93. doi: 10.1097/MOO.0000000000000079. PMID 25188429
- [Background] Kujawa SG, Liberman MC. Adding insult to injury: cochlear nerve degeneration after "temporary" noise-induced hearing loss. J Neurosci. 2009 Nov 11;29(45):14077-85. doi: 10.1523/JNEUROSCI.2845-09.2009. PMID 19906956
- [Background] Lin HW, Furman AC, Kujawa SG, Liberman MC. Primary neural degeneration in the Guinea pig cochlea after reversible noise-induced threshold shift. J Assoc Res Otolaryngol. 2011 Oct;12(5):605-16. doi: 10.1007/s10162-011-0277-0. Epub 2011 Jun 18. PMID 21688060
- [Background] Snapp HA, Vanlooy L, Kuzbyt B, Kolberg C, Laffitte-Lopez D, Rajguru S. Peripheral vestibular loss in noise-exposed firefighters. Front Integr Neurosci. 2023 Oct 2;17:1236661. doi: 10.3389/fnint.2023.1236661. eCollection 2023. PMID 37849955
- [Background] Williams EC, Ma Y, Loo DM, Schaefer Solle N, Millet B, Harris K, Snapp HA, Rajguru SM. Monitoring Occupational Noise Exposure in Firefighters Using the Apple Watch. Int J Environ Res Public Health. 2023 Jan 28;20(3):2315. doi: 10.3390/ijerph20032315. PMID 36767682
- [Background] Snapp HA, Schaefer Solle N, Millet B, Rajguru SM. Subclinical Hearing Deficits in Noise-Exposed Firefighters. Int J Environ Res Public Health. 2022 Sep 3;19(17):11028. doi: 10.3390/ijerph191711028. PMID 36078744
- [Background] Snapp HA, Millet B, Schaefer-Solle N, Rajguru SM, Ausili SA. The effects of hearing protection devices on spatial awareness in complex listening environments. PLoS One. 2023 Jan 12;18(1):e0280240. doi: 10.1371/journal.pone.0280240. eCollection 2023. PMID 36634110
- [Background] Snapp HA, Coto J, Solle NS, Khan U, Millet B, Rajguru SM. Risk-taking propensity as a risk factor for noise-induced hearing loss in the general population. Int J Audiol. 2023 Dec;62(12):1166-1175. doi: 10.1080/14992027.2022.2114023. Epub 2022 Sep 1. PMID 36047290
- [Background] Millet B, Snapp HA, Rajguru SM, Schaefer Solle N. Prevalence of Hearing Loss and Perceptions of Hearing Health and Protection among Florida Firefighters. Int J Environ Res Public Health. 2023 Feb 21;20(5):3826. doi: 10.3390/ijerph20053826. PMID 36900832
- [Background] Tamames I, King C, Bas E, Dietrich WD, Telischi F, Rajguru SM. A cool approach to reducing electrode-induced trauma: Localized therapeutic hypothermia conserves residual hearing in cochlear implantation. Hear Res. 2016 Sep;339:32-9. doi: 10.1016/j.heares.2016.05.015. Epub 2016 May 31. PMID 27260269
- [Background] Singh J, Barrett J, Sangaletti R, Dietrich WD, Rajguru SM. Additive Protective Effects of Delayed Mild Therapeutic Hypothermia and Antioxidants on PC12 Cells Exposed to Oxidative Stress. Ther Hypothermia Temp Manag. 2021 Jun;11(2):77-87. doi: 10.1089/ther.2019.0034. Epub 2020 Apr 17. PMID 32302519
- [Background] Sangaletti R, Tamames I, Yahn SL, Choi JS, Lee JK, King C, Rajguru SM. Mild therapeutic hypothermia protects against inflammatory and proapoptotic processes in the rat model of cochlear implant trauma. Hear Res. 2023 Feb;428:108680. doi: 10.1016/j.heares.2022.108680. Epub 2022 Dec 20. PMID 36586170
- [Background] Patel J, Szczupak M, Rajguru S, Balaban C, Hoffer ME. Inner Ear Therapeutics: An Overview of Middle Ear Delivery. Front Cell Neurosci. 2019 Jun 11;13:261. doi: 10.3389/fncel.2019.00261. eCollection 2019. PMID 31244616
- [Background] Eshraghi AA, Nazarian R, Telischi FF, Rajguru SM, Truy E, Gupta C. The cochlear implant: historical aspects and future prospects. Anat Rec (Hoboken). 2012 Nov;295(11):1967-80. doi: 10.1002/ar.22580. Epub 2012 Oct 8. PMID 23044644